CLINICAL TRIAL: NCT03486054
Title: A Randomized, Controlled, Phase I Clinical Trial to Assess the Safety of Whole Blood Treated With Amustaline (S-303) and Glutathione (GSH), a Pathogen Reduction System in Anemic Patients.
Brief Title: INTERCEPT Safety Evaluation in Anemic Patients
Acronym: POINT1africa
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: strategic reasons
Sponsor: Swiss Transfusion SRC (Other)
Collaborators: Cerus Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 702005
Record Dates: First submitted 2018-03-06; First posted 2018-04-03 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Anemia
Keywords: Anemia; Transfusion; Pathogen inactivation; low-resource; Sub-saharan Africa; Côte d'Ivoire; Transfusion-transmitted infection; Red Blood Cells; Whole blood; Pathogen reduction
MeSH Terms: conditions — Anemia; Transfusion Reaction

STUDY DESIGN:
Intervention Model Description: Experimental Arm: INTERCEPT Treated Whole Blood Control Arm: Standard of Care (Red Blood Cells, Whole Blood)
Masking Description: Randomized, controlled, open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm A (Experimental): Whole blood treated with amustaline and glutathione, a pathogen reduction technology (PRT), ordered and administered to study patients by their treating physicians
  Interventions: Device: INTERCEPT
- Control Arm B (Active Comparator): Standard of Care (either red blood cells or whole blood)
  Interventions: Device: Standard of Care

INTERVENTIONS:
Device: INTERCEPT — The pathogen reduction process begins with a unit of whole blood collected according to local standards and procedures at the blood center. The blood unit is treated with amustaline and glutathione (INTERCEPT blood system for whole blood) according to manufacturer's instructions. The INTERCEPT blood system is performed on a single unit of not leuco-reduced whole blood treated with amustaline and glutathione in CPD
  Other Names: Experimental
  Arms: Experimental Arm A
Device: Standard of Care — The control article is Standard of Care, either RBC or whole blood collected by the Centre National de Transfusion Sanguine (CNTS), processed according to the local procedure and in compliance with quality criteria defined by the manufacture regarding the volume, hemoglobin content, hematocrit, storage temperature, age of blood and storage in the predefined anticoagulant solution.
  Other Names: Control
  Arms: Control Arm B

SUMMARY:
The pathogen reduction (PR) system for Whole Blood (WB) using Amustaline (S-303) and Glutathione (GSH) has a potential to decrease transfusion-transmitted infection. There is scientific basis to hypothesize, that cells containing DNA and RNA such as bacteria, viruses and parasites that could be present in blood collected from asymptomatic infected donors are inactivated in the treated whole blood and therefore reduce the risk of transfusion-transmitted infections. The aim of the study is to gather data to support the safety of whole blood products that underwent treatment with amustaline and glutathione and data to support a larger sufficiently powered efficacy study. This study will evaluate the safety of the system for whole blood in adult patients with anemia.

This study is designed as a randomized, controlled, open-label study. The aim is to explore the safety of the whole blood product treated with a PR system using amustaline and glutathione.

The study will enroll 20 patients with anemia. 20 patients will be randomized either to treated WB (Test) or Standard of Care, either Red Blood Cells or Whole Blood (Control).

DETAILED DESCRIPTION:
Screening:

All potentially eligible patients at the participating institution will be approached for study consent prior to study transfusion. Enrolled patients will be asked for consent to the storage of their samples for a future project in TTI Project. Illiterate patients can be consented by an impartial witness.

Patients who consent to the study will be assigned a study ID number and undergo screening.

Screening data collection and procedures will include: Demographics (age, sex), vital signs, height, weight, indication for anticipated transfusion, medical history including history of bleeding and transfusion and concomitant medications. A physical examination, including skin inspection, will be performed. Blood samples will be drawn for a hematological panel (including complete blood count, blood chemistry, blood type, coagulation (aPTT, PT and/or INR) and pregnancy test (if applicable). Immunohematology tests will be performed in a patient's sample at the blood transfusion center. This includes the Direct Antibody Test (DAT), immune reactivity to RBCs that have been processed with the INTERCEPT Blood System (IBS RBC), red cell alloantibody screen (Indirect Antibody Test (IAT) / Indirect Coombs).

Blood samples (pre/post-treatment) for future research on transfusion-transmitted infections will be archived in a biobank of the Institut Pasteur de Côte d'Ivoire (IPCI)

Randomization:

After successful screening, eligible patients will be assigned to a treatment arm by randomization. Randomization will be performed in the blood center by sequentially selecting a randomization envelope starting with the lowest number (e.g., 1 for the first eligible subject in ascending order up to envelope number 20 for the 20th subject).

The ratio of patients assigned to the Test and Control group will be 1:1. Each subject will receive a Test product or SOC. The assigned blood product number must be noted on the randomization assignment envelope and on the release form. The product number will also be entered into the case report form (CRF).

The replacement strategy in this Phase I clinical trial is based on the aim to reach twenty evaluable patients ("evaluable patients" is defined as those patients who are randomized and receive any study transfusion).

If a randomized subject withdraws or is withdrawn from the study prior to the administration of any study transfusion, or does not receive any study transfusion through 7-days post-randomization, this subject will be replaced by the next eligible subject using the same randomization envelope. If a randomized subject receives a conventional (untreated) blood transfusion prior to study transfusion, the patient will be replaced as described above.

All patients who received at least one study product will be included into the analysis of evaluable patients and followed up to the final study visit on Day 58.

All used and unused randomization envelopes will be kept in the Site File for reconciliation.

Pre-transfusion visit:

Vital signs, height, weight, hemoglobin will be assessed and urine dipstick test for detection of blood will be performed. If the patient consented to future research on TTI, a sample is drawn.

Treatment:

Patients will be transfused with one investigational product or SOC on Day 1. In case he or she requires further transfusion support to treat anemia, enrolled patients may be treated with a second study transfusion. A patient who requires a second blood component will receive a second treatment with a study product from the assigned treatment arm. This patient will be included into the analysis of evaluable patients and followed up to Day 58, the end of study visit.

Post-transfusion visit(s):

Patients will be hospitalized for 24 hours after each study transfusion to allow close monitoring and data collection uniquely for the study purpose since their condition would allow an outpatient treatment. 3 hours and 6 hours after initiating each study transfusion vital signs, skin inspection, and urine dipstick will be performed.

24-hours post-transfusion vital signs, concomitant medication/intervention will be assessed, laboratory samples for hemoglobin, coagulation assays (aPTT, PT and/or INR) and potassium and a sample for determination of residual S-300 will be taken.

If a subject consented to future research on TTI, a second blood sample (post-transfusion) will be taken and archived in the biobank.

In case clinical symptoms of transfusion-related bacterial contamination occur, a blood sample will be taken during the post-transfusion period and sent for microbiological analysis. Those patients will be treated according to local SOC.

Safety Follow-up visit Day 28 (+/-3 days after last study transfusion):

At day 28 (+/-3 days) a physical examination, vitals and blood samples will be collected for laboratory analysis of safety variables (e.g., complete blood count, coagulation, blood chemistry) and urine dipstick.

All Adverse Events (AE), Transfusion Reactions (TR) and unanticipated adverse device effects will be reviewed and recorded for the period from the first study transfusion through day 28 after the last study transfusion.

The Investigators will assess each AE/TR for relation to the study transfusion. Available clinical diagnostic tools will be used to classify occurring transfusion reactions by the definitions of Swissmedic grading scale.

Final study visit Day 58 (+/-7 days after last study transfusion) At the final study visit, the immune reactivity of patient serum to RBCs treated with amustaline/GSH and a DAT test will be performed.

SAEs will be reviewed and recorded for the period of 58 days up to the final study visit.

The Investigators will assess each Serious Adverse Event (SAE) for relation to the study transfusion. Depending on the availability of clinical diagnostic tools, the transfusion reactions will be classified by the definitions of Swissmedic grading scale.

ELIGIBILITY:
Stable anemic patients according to local clinical guidelines qualified to receive a whole blood transfusion in a non-emergency situation.

Inclusion criteria:

Patients must fulfill all of the following inclusion criteria:

1. Patients must be18 years of age or older;
2. Patients must have a hemoglobin level of >/= 5.0 g/dl. Patients with hemoglobin levels of >7.0 will not be excluded provided the patient's physician deems transfusion is needed to address anemia-induced symptoms.
3. Patients must sign informed consent prior to initiation of any study-specific procedure / treatment. Enrolled patients may give additional consent for specimens collected during this study to be used for future research on TTI. Patients may participate in the main trial and decline collection of specimens for future research on TTI.
4. Patients must agree to be hospitalized for a maximum of 72 hours after initiation of a study transfusion;
5. Female patients of childbearing potential must:

   1. have a negative serum pregnancy test within 72 hours prior to receiving the first study blood to rule out pregnancy, and
   2. use at least one method of birth control that results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly. These include combined oral contraceptives, implants, injectable, some intrauterine devices, sexual abstinence or vasectomized partner. The selected method must be used for the duration of study participation that means from day 1 (day of initiation of study transfusion) until day 58 (Final Study Visit).

Exclusion criteria:

The presence of any one of the following exclusion criteria will lead to exclusion:

Stable anemic patients according to local clinical guidelines qualified to receive a transfusion in a non-emergency situation.

Inclusion criteria:

Patients must fulfill all of the following inclusion criteria:

1. Patients must be18 years of age or older;
2. Patients must have a hemoglobin level of >/= 5.0 g/dl. Patients with hemoglobin levels of >7.0 will not be excluded provided the patient's physician deems transfusion is needed to address anemia-induced symptoms.
3. Patients must sign informed consent prior to initiation of any study-specific procedure / treatment. Enrolled patients may give additional consent for specimens collected during this study to be used for future research on TTI. Patients may participate in the main trial and decline collection of specimens for future research on TTI.
4. Patients must agree to be hospitalized for a maximum of 72 hours after initiation of a study transfusion;
5. Female patients of childbearing potential must:

   1. have a negative serum pregnancy test within 72 hours prior to receiving the first study blood to rule out pregnancy, and
   2. use at least one method of birth control that results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly. These include combined oral contraceptives, implants, injectable, some intrauterine devices, sexual abstinence or vasectomized partner. The selected method must be used for the duration of study participation that means from day 1 (day of initiation of study transfusion) until day 58 (Final Study Visit).

Exclusion criteria:

The presence of any one of the following exclusion criteria will lead to exclusion:

1. Patients with blood group AB (due to concern of limited supply).
2. Positive antibody screening reaction specific to red blood cells treated by amustaline and glutathione (GSH).
3. Positive red cell alloantibody screening (IAT) / presence of red cell antibodies;
4. Patient has ongoing clinical-significant bleeding described as grade 2 or more according to CTCAE v5.0.
5. Lifelong history of major bleeding due to congenital or acquired coagulopathy.
6. History of thrombosis or thromboembolic events.
7. Blood in urine or feces in the last 30 days.
8. Pre-transfusion thrombocyte counts of < than 50 Giga/l (x109).
9. Oral, intravenous or sub-cutaneous prophylactic or therapeutic anticoagulants.
10. Central body temperature increase of ≥ 2 °C within 24 hours before transfusion.
11. Clinical signs of ongoing sepsis including fever > 39°C with signs of a systemic, inflammatory response.
12. Abnormal activated partial thromboplastin time (aPTT) and/or abnormal prothrombin time (PT) or INR laboratory results
13. Transfusion of a blood product within 2 weeks prior to enrollment.
14. Abnormal total bilirubin (2 x upper limit of normal) levels and /or clinical signs of jaundice.
15. Previous treatment with other pathogen-reduced blood products.
16. Sickle cell anemia.
17. Malignant cancer patients having received chemotherapy within 12 months.
18. Patients in need of multiple RBC or WB transfusions in the first 24 hours according to the attending physician's judgment (i.e., more than one product).
19. Pregnant or breast feeding.
20. Inability to comply with the protocol in the opinion of the investigator.
21. Participation in any other type of clinical study either concurrently or within the previous 30 days: investigational blood products, nutrition, pharmacologic agents or imaging materials, including dyes, investigational surgical techniques, or devices (studies of psychology or socioeconomic issues are not grounds for exclusion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Severe Transfusion Reactions | 24 hours
  The primary safety outcome will be assessed by the occurrence of transfusion reactions >= grade 2 according to the Swissmedic transfusion reaction grading and causality criteria (Appendix 1), during the first 24 hours following administration of each study transfusion, with probable, possible or certain causality to the transfused product

SECONDARY OUTCOMES:
Adverse events | 58 (+/-7)
  All adverse events including all transfusion reactions within 28 (+/-3) days and all SAEs within 58 (+/- 7) days after last study transfusion.
Treatment-emergent antibodies | 58 (+/-7)
  Treatment-induced antibodies to amustaline/GSH treated RBCs within 58 (+/-7) days after last study transfusion
Treatment-emergent auto-antibodies | 58 (+/-7)
  Treatment emergent auto-antibody within 58 (+/-7) days after study transfusion
Hemoglobin increment | 24 hours
  The hemoglobin increment 24h post transfusion will be calculated as the difference between the hemoglobin value most proximate before the transfusion and approximately 24h post transfusion, adjusted by hemoglobin content transfused.

CONTACTS AND LOCATIONS:
Overall Officials: Soraya Amar, MD, Study Director — Transfusion SRC

IPD SHARING:
Plan to Share IPD: No